CLINICAL TRIAL: NCT03882840
Title: Induced-T Cell Like NK Cellular Immunotherapy for Cancers That Are Lack of MHC-I Expression
Brief Title: Induced-T Cell Like NK Cellular Immunotherapy for Cancer Lack of MHC-I
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Hunan Zhaotai Yongren Medical Innovation Co. Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZZITNK-007
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Anti-cancer Cell Immunotherapy; T Cell and NK Cell
Keywords: Solid Tumor, ITNK, CAR-ITNK

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ITNK cell therapy group (Experimental): Patient-originated and induced T-to-natural killer (ITNK) cells, will be administrated to kill tumor cells.
  Interventions: Biological: ITNK cell therapy
- CAR-ITNK cell therapy group (Experimental): Patient-originated and induced T-to-natural killer (ITNK) cells with CAR-engineered, will be administrated to kill tumor cells.
  Interventions: Biological: ITNK cell therapy

INTERVENTIONS:
Biological: ITNK cell therapy — Infusion of ITNK/CAR-ITNK cells

SUMMARY:
T effector cells and NK cells have mutual compensatory killing functions on various of cancer types. For those cancers that have no available targets for CAR-T cell generations, we established potent T cell-like NK cells (ITNK) with a specific conversion protocol for the T cells from the patient, to perform anti-cancer therapy, especially for those cancers that are lack of MHC-I molecule expression. We have finished pre-clinical investigations for the ITNK or CAR-ITNK cell therapy and scheduled to start a clinical phase I study.

DETAILED DESCRIPTION:
One gene can be knockout of the T cells to produce a T-like NK cells which obtain killing function of both T effector cells and NK cells. We will collect appropriate patient's T cells, produce T-like NK cells (ITNK), and infuse the ITNK/CAR-ITNK cells back to the patients to treat various of cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced cancer, which express low or no MHC-I.
2. Life expectancy >12 weeks
3. Adequate heart,lung,liver,kidney function
4. Available autologous T cells
5. Informed consent explained to, understood by and signed by patient/guardian. 6. Patient/guardian given copy of informed consent.

Exclusion Criteria:

1. Had accepted gene therapy before;
2. Severe virus infection such as HBV,HCV,HIV,et al
3. Known HIV positivity
4. History of liver or other organ transplantation
5. Active infectious disease related to bacteria, virus,fungi,et al
6. Other severe diseases that the investigators consider not appropriate;
7. Pregnant or lactating women
8. Systemic steroid treatment (greater than or equal to 0.5 mg prednisone equivalent/kg/day)
9. Other conditions that the investigators consider not appropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
The safety and tolerance of the ITNK cell immunotherapy | 2 years
  A dose limiting toxicity is defined as any toxicity that is considered to be primarily related to the ITNK cells, which is irreversible, or life threatening or hematologic or non-hematologic Grade 3-5. Incidence of treatment-emergent adverse events will be calculated as standard methods.

SECONDARY OUTCOMES:
Percent of Patients with best response as either complete remission or partial remission. | 2 years
  Response rates will be estimated as the percent of patients whose best response is either complete remission or partial remission by combining the data from the patients. To compare with historical data, a 95% confidence interval will be calculated for the response rate.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD, PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Li P, Burke S, Wang J, Chen X, Ortiz M, Lee SC, Lu D, Campos L, Goulding D, Ng BL, Dougan G, Huntly B, Gottgens B, Jenkins NA, Copeland NG, Colucci F, Liu P. Reprogramming of T cells to natural killer-like cells upon Bcl11b deletion. Science. 2010 Jul 2;329(5987):85-9. doi: 10.1126/science.1188063. Epub 2010 Jun 10. PMID 20538915
- [Derived] Jiang Z, Qin L, Tang Y, Liao R, Shi J, He B, Li S, Zheng D, Cui Y, Wu Q, Long Y, Yao Y, Wei Z, Hong Q, Wu Y, Mai Y, Gou S, Li X, Weinkove R, Norton S, Luo W, Feng W, Zhou H, Liu Q, Chen J, Lai L, Chen X, Pei D, Graf T, Liu X, Li Y, Liu P, Zhang Z, Li P. Human induced-T-to-natural killer cells have potent anti-tumour activities. Biomark Res. 2022 Mar 24;10(1):13. doi: 10.1186/s40364-022-00358-4. PMID 35331335